CLINICAL TRIAL: NCT05259124
Title: The Ability of Perfusion Index and Positional Perfusion Index Variation to Predict Spinal Anesthesia-induced Hypotension in Elderly Patients: A Prospective Observational Study
Brief Title: The Ability of Perfusion Index and Positional Perfusion Index Variation to Predict Spinal Anesthesia-induced Hypotension in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud AbdelKader, principal investigator, Cairo University
Other Study IDs: N-122-2021
Record Dates: First submitted 2022-01-17; First posted 2022-02-28 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Spinal Anesthesia Induced Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: positional perfusion index variation — positional perfusion index variation to predict spinal anesthesia-induced hypotension in elderly patients

SUMMARY:
In this study, we will test the ability of positional perfusion index variation to predict post-spinal anesthesia hypotension in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or more.
* ASA score I & II.
* Patients scheduled for surgeries under spinal anesthesia.

Exclusion Criteria:

* Negative consent.
* pre-existing hypertension
* Diabetes mellitus or autonomic neuropathy.
* Emergency operations.
* Absolute contraindications or failure to perform spinal anesthesia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A total of 68 consecutive elderly patients, aged >65 years scheduled for elective surgical operations under spinal anesthesia will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
The sensitivity of perfusion index postural change in predicting spinal anesthesia-induced hypotension in elderly patients. | 30 minutes after spinal anesthesia
  The sensitivity of incremental change of a measured perfusion index pre and post spinal anesthesia

SECONDARY OUTCOMES:
incidence of spinal anesthesia induced hypotension in elderly | 30 minutes after spinal anesthesia
  incidence of spinal anesthesia induced hypotension in elderly
• The sensitivity of supine perfusion index to predict spinal anesthesia-induced hypotension in elderly patients. | 30 minutes after spinal anesthesia
  • The sensitivity of supine perfusion index to predict spinal anesthesia-induced hypotension in elderly patients.
• The sensitivity of sitting perfusion index to predict spinal anesthesia-induced hypotension in elderly patients. | 30 minutes after spinal anesthesia
  • The sensitivity of sitting perfusion index to predict spinal anesthesia-induced hypotension in elderly patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospital, Cairo, Giza Governorate, Egypt